CLINICAL TRIAL: NCT06081647
Title: The Efficacy and Safety of the COMBO Endoscopy Oropharyngeal Airway Reduce the Incidence of Hypoxia in Patients Undergoing Gastrointestinal Endoscopy Sedated With Propofol.
Brief Title: The Efficacy and Safety of the COMBO Endoscopy Oropharyngeal Airway in Gastrointestinal Endoscopy Procedure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, diansan su, Vice Chair of the Department of Anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LY2023-159-B
Record Dates: First submitted 2023-09-19; First posted 2023-10-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hypoxia; Gastric Polyp; Colon Cancer; Esophageal Cancer
Keywords: the COMBO Endoscopy Oropharyngeal Airway; Hypoxia; Gastrointestinal Endoscopy; Propofol; Sedation
MeSH Terms: conditions — Hypoxia; Polyposis, Gastric; Colonic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the COMBO Endoscopy Oropharyngeal Airway Group (Experimental): In this group, patients use the COMBO Endoscopy Oropharyngeal Airway for oxygenation.
  Interventions: Device: the COMBO Endoscopy Oropharyngeal Airway
- Regular Nasal Cannula Group (Active Comparator): In this group, patients use the regular nasal cannula for oxygenation.
  Interventions: Device: Regular Nasal Cannula

INTERVENTIONS:
Device: the COMBO Endoscopy Oropharyngeal Airway — Using the COMBO Endoscopy Oropharyngeal Airway for oxygenation.
  Arms: the COMBO Endoscopy Oropharyngeal Airway Group
Device: Regular Nasal Cannula — Using regular nasal cannula for oxygenation.
  Arms: Regular Nasal Cannula Group

SUMMARY:
Hypoxia represents the prevailing adverse occurrence during the sedation of patients undergoing gastrointestinal endoscopy with propofol. A recent innovation in this domain is the COMBO Endoscopy Oropharyngeal Airway-a multifaceted device that encompasses capnography monitoring, bite block , oxygenation support, and oropharyngeal airway management. This device has been purposefully designed to cater to the unique requirements of endoscopic procedures. The principal objective of our randomized study is to assess the efficacy and safety of the COMBO Endoscopy Oropharyngeal Airway reduce the incidence of hypoxia on patients undergoing gastrointestinal endoscopy under propofol sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18≤ Age ≤60.
* Patients undergoing gastroendoscopy and/or colonoscopy procedure.
* Patients have signed the informed consent form.
* The ASA classification ranges from I to II.
* The estimated duration of the procedure does not exceed 45 minutes.

Exclusion Criteria:

* Patients who exhibit contraindications to oropharyngeal airway ventilation, such as coagulation disorders, a predisposition to oral and nasal bleeding, mucosal damage, or anatomical constraints impeding oropharyngeal channel placement.
* Severe cardiac insufficiency, defined as a maximal exercise capacity of less than 4 metabolic equivalents (METs).
* Profound renal insufficiency necessitating preoperative dialysis.
* A confirmed severe liver dysfunction.
* Patients diagnosed with chronic obstructive pulmonary disease (COPD) or those presently experiencing other acute and chronic pulmonary conditions necessitating prolonged or intermittent oxygen therapy.
* Elevated intracranial pressure.
* Upper respiratory tract infections, encompassing the oral, nasal, and pharyngeal regions.
* Fever, defined as a core body temperature exceeding 37.5 degrees Celsius.
* Pregnancy or lactation.
* Hypersensitivity reactions to sedatives like propofol or medical equipment such as adhesive tape.
* Urgent surgical intervention.
* Polytrauma.
* Peripheral oxygen saturation (SpO2) levels below 95% while breathing room air preoperatively.
* BMI<18.5 or BMI>30.
* Patients with a documented history of substance abuse, specifically drugs and/or alcohol, within the two years preceding the commencement of the screening period. Substance abuse in this context is defined as consuming more than three standard alcoholic beverages daily, roughly equivalent to 10g of alcohol or 50g of Chinese Baijiu.
* Patients with a history of mental and neurological disorders, including but not limited to depression, severe central nervous system depression, Parkinson's disease, basal ganglia lesions, schizophrenia, epilepsy, Alzheimer's disease, and myasthenia gravis.
* Presently engaged in concurrent participation in additional clinical trials.
* Patients considered ineligible by researchers for inclusion in this clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  (75% ≤ SpO2 < 90% for <60 s)

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  (90% ≤ SpO2 < 95%)
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  (SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s)

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Shangdong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai, Shanghai Municipality
  - Tongji Hospital Of Tongji University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affliated To Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghia
  - The First Affliated Hospital of Xi'an Jiangtong University, Xi’an, Shanxi
  - Tianjin Mediacal University General Hospital, Tianjin, Tianjin Municipality
  - The First Affliated Hospital, Zhejiang University School Of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data (including data dictionaries) and analysis codes generated in this study are available upon reasonable request. Additional documents, such as the study protocol and statistical analysis plan, can also be provided. Data will be accessible beginning 3 months after article publication for at least 5 years. Researchers seeking access must submit a request to the corresponding author for approval, which will be granted based on scientific merit and compliance with a data sharing agreement.

REFERENCES:
- [Derived] Zhang Y, Shi M, Qu Y, Cheng X, Zhang J, Guo S, Zheng Y, Su D. Efficacy and safety of the COMBO endoscopy oropharyngeal airway in gastrointestinal endoscopy: a study protocol for a multicenter randomized controlled trial. Trials. 2025 Dec 13. doi: 10.1186/s13063-025-09351-2. Online ahead of print. PMID 41390738